CLINICAL TRIAL: NCT01802957
Title: Health Facility Networking for Maternal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Maternal Health Task Force (Unknown); St. Paul's Hospital Millennium Medical College, Ethiopia (Other); Addis Continental Institute of Public Health (Other); Institute for Clinical Effectiveness and Health Policy (Other)
Responsible Party: Principal Investigator, Ana Langer, Professor of the Practice of Public Health Coordinator of the Dean's Special Initiative in Women and Health, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MHTF IR Ethiopia
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Provider Skill; Provider Confidence; Maternal Health; Referral Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- St. Paul and Networked Health Centers (Other): An uncontrolled before and after design with baseline and follow-up cross sectional measurements will be used at the overall site level (St. Paul Hospital and the 8 associated HCs). There will be no control unit.
  Interventions: Other: Training of health workers in Basic Obstetric Emergency Care; Other: Hospital-health center networking system; Other: Post Basic Emergency Obstetric Training Mentorship; Other: Team-Based Supportive supervision; Other: Midwives exchange program; Other: Strengthening the referral network; Other: Facility Checklists; Other: Emergency Drills

INTERVENTIONS:
Other: Training of health workers in Basic Obstetric Emergency Care — Health workers at the eight health centers will be trained in maternal, newborn, and child health (MNCH) care, including all basic emergency obstetric and neonatal care (BEmONC) signal functions and other essential MNCH services. The training is a three week competency-based curriculum developed recently by the Ethiopian Federal Ministry of Health (FMoH).
Other: Hospital-health center networking system — A key intervention will be the creation of an effective, formalized networking system between Saint Paul Millennium Hospital and its eight satellite health centers in Addis Ababa. The networking system will create a conducive environment for the transfer of knowledge and skills between health care providers working at the hospital and in the health centers. Monthly review meetings will bring together staff from the hospital and health centers, and dedicated cell phones will be distributed to improve communication between the networked facilities.
Other: Post Basic Emergency Obstetric Training Mentorship — At Saint Paul Millennium Hospital and the health centers, providers who have undergone BEmONC training will undergo regular monthly mentorship visits for the first six months post training. The frequency of visits after six months will be adjusted based on the retention of BEmONC skills and provider performance
Other: Team-Based Supportive supervision — Saint Paul Hospital will use team-based models to provide supportive supervision to health centers in its network. Representatives of the supportive supervision teams may, in addition to Saint Paul Hospital employees, include representatives from the Addis Ababa Regional Health Bureau.
Other: Midwives exchange program — Saint Paul Millennium Hospital's maternity wards are often over-crowded and have to turn patients away. Health professionals incorrectly refer non-complicated deliveries, resulting in the occupation of beds that should be used for emergency deliveries. This action is attributed to inexperienced midwives at the health center level who are uncomfortable performing normal labor and delivery duties. In order to address this challenge, this project will establish an exchange program in which well-trained, experienced midwives from the hospitals will temporarily exchange places with less-experienced midwives in the health centers. This exchange would allow less-experienced midwives to work in the hospital environment, gaining the experience and confidence necessary to attend normal deliveries and identify appropriate referrals.
Other: Strengthening the referral network — Mechanisms and protocols for smooth communication between the health centers and the hospital have been developed, allowing health centers to utilize the hospital's ambulance, and implementing mechanisms for back referrals and feedback. To facilitate this work, we will support the use of dedicated cell phones in each of the eight networked facilities and at Saint Paul Millennium Hospital, and institute referral log books at both the referring and receiving institutions.
Other: Facility Checklists — Facility checklists will be used daily in each of the facilities to assess readiness for obstetric emergencies. Formally, the checklists will be used at the quarterly supportive supervision visits, to assess improvements over time.
Other: Emergency Drills — Non-punitive obstetric drills will provide multiple measurable indicators of quality maternal care, will illustrate opportunities for improving facility capabilities and provider care, and will allow providers to assess appropriate referral mechanisms and facility readiness. Incorporating emergency drills into current training and at all levels of health facilities will also give providers hands-on experience

SUMMARY:
This study will introduce a multi-faceted intervention package which will be implemented in the newly developed network of St. Paul's Hospital Millennium Medical College (St. Paul) and the surrounding seven satellite health centers. The goal is to assess if this group of interventions improve the skills and confidence of providers to handle obstetric emergencies, if they streamline the referral process and if they result in improved maternal/newborn health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Sample population for each data collection instrument:

Baseline/Endline:

Key Informant Interviews:

* St. Paul hospital: Maternal Child Health (MCH) Head, Midwife/nurse from Labor and Delivery (L&D), Midwife/nurse from Emergency
* Health Centers: Medical Director, Head of MCH (midwife) Midwife from L&D, Referral focal person

Health Facility Assessment:

- Manager/most senior health worker asked (one from each facility)

Provider Survey:

- All providers in the MCH at both the hospital and health center level

Chart review:

- All deliveries in all centers will be screened during the intervention phase. Data on every birth will be collected from the log books of each facility. The data collector will then find the medical record of that patient to assess the Standard of Care (SOC) during Ante-natal care (ANC)- if available from the chart, L&D and screen for an obstetric complication. If there was a complication, the near miss data will be collected.

Telephone registration log book:

- all phone calls between HC and Hospital

Facility Checklists:

- Forms completed by Supportive Supervision Teams at quarterly visits

Standardized BEmONC training evaluation

- Will be given to every provider undergoing the training, as part of the training curriculum.

Monthly mentoring evaluations - for the six months post-training mentorship, for all providers who have undergone BEmONC training.

Supportive Supervision Gap Identification Checklists

- Collected quarterly from each of the 9 facilities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10787 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improved provider skill levels | One Year
  Provider skill will be measured through baseline and endline evaluations, mentoring reports, and the standardized evaluations used in the Basic Emergency Obstetric Care trainings.
Improved provider self-efficacy | One Year
  Improved provider confidence will be assessed at baseline and at endline with a standardized data collection instrument.
Increased use of effective interventions for obstetric emergencies | One Year
  Continuous data extraction from patient charts will be used to assess the appropriate treatment for obstetric emergencies over the study period. Additionally changes in time-to-treatment for post-partum hemorrhage and pre-eclampsia/eclampsia cases will also be assessed from patient charts.
Improved standards of care for pregnant women | One Year
  Continuous extraction from patient records throughout the study period will be used to assess the trends in the Standards of Care (SOC) for Ante-natal (ANC), and care during Labor and Delivery.
Improved Referral Systems | One Year
  * Decreases the proportion of referrals made without proper prior communication to the receiving health facility
  * Formalized feedback mechanisms between Saint Paul and the Health Centers
  * Decreased number of inappropriate referrals from Health Centers to St. Paul
  * Appropriate back-referrals from St. Paul to Health Centers
  Data on Health Center/Hospital communication and referrals will be collected through phone logs, and referral sheets.

SECONDARY OUTCOMES:
Sustainable, continuous quality improvement cycles through supportive supervision | One year
  Quarterly, a supportive supervision team will visit each of the health facilities involved in this study, and, using a checklist and a participatory approach, will identify areas to improve the quality of care provided. Each action item will will have a person assigned to it, and a plan to resolve the issue. Follow up supportive supervision visits will begin with an assessment of the previous visit's action plan, and then work to identify new areas for quality improvement. This process is iterative.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Langer, MD, Principal Investigator — Harvard School of Public Health (HSPH); Yemane Berhane, MD, MPH, PhD, Principal Investigator — Addis Continental Institute of Public Health; Delayehu Bekele, MD, Principal Investigator — St. Paul's Hospital Millennium Medical College, Ethiopia; Fernando Althabe, MD, Study Director — Institute for Clinical Effectiveness and Health Policy
Locations (8):
- Ethiopia (8):
  - Addis Ketema Health Center, Addis Ketema Subcity, Woreda 4
  - Woreda 7 Health Center, Addis Ketema Subcity, Woreda 9, Addis Ababa,
  - Semen Health Center, Arada Sub City, Addis Ababa
  - Selam Health Center, Gulele Sub City, Woreda 9, Addis Ababa
  - St. Paul Hospital Millennium Medical College, Gulele Subcity, Addis Ababa
  - Shegole Health Center, Gulele Subcity, Woreda 10, Addis Ababa
  - Woreda 7 Health Center, Gulele Subcity, Woreda 7
  - Kolfe Health center, Kolfe Sub City, Woreda 2, Addis Ababa